CLINICAL TRIAL: NCT01821209
Title: A Randomized Study of Intra-operative Autologous Retropubic Urethral Sling on Urinary Control After Robot Assisted Radical Prostatectomy
Brief Title: A Study of Intra-operative Autologous Retropubic Urethral Sling on Urinary Control After Robot Assisted Radical Prostatectomy
Acronym: Sling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SLING2013
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Men With Prostate Cancer Undergoing Robot Assisted Radical Prostatectomy
Keywords: prostate cancer, robotic surgery, urethral sling,
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Standard robot assisted radical prostatectomy
- Sling (Experimental): Placement of sling at time of robot assisted radical prostatectomy
  Interventions: Procedure: Placement of sling

INTERVENTIONS:
Procedure: Placement of sling — Placement of a retropubic urethral sling will involve dissection and harvesting of the right and left vas deferens, which we will be taken out of the body by the bed side assistant who will suture the two vas deferens together in a side to side fashion with the smaller of the two vas deferens placed in the middle of the larger one. A single 3-0 V-lock suture on a CV23 needle will be placed through one end of the vas sling and then passed into the body by the bed side assistant. The sling will then be placed on the rectum below the site of the vesicourethral anastamosis and the anastamosis will be completed. The sling will then be placed around the vesicourethral anastomosis, suspended to the pubic symphysis and tensioned to allow elevation of the vesicourethral anastomosis.
  Arms: Sling

SUMMARY:
Placement of an autologous retropubic urethral sling at the time of robot assisted radical prostatectomy will improve the recovery of continence after radical prostatectomy

DETAILED DESCRIPTION:
This is a phase 2 single blinded study of patients undergoing robot assisted radical prostatectomy who are randomized to placement of an autologous retropubic urethral sling or not. Placement of a retropubic urethral sling will involve dissection and harvesting of the right and left vas deferens, which will be taken out of the body by the bed side assistant who will suture the two vas deferens together in a side to side fashion with the smaller of the two vas deferens placed in the middle of the larger one. A single 3-0 V-lock suture on a CV23 needle will be placed through one end of the vas sling and then passed into the body by the bed side assistant. The sling will then be placed on the rectum below the site of the vesicourethral anastamosis and the anastamosis will be completed. The sling will then be placed around the vesicourethral anastomosis, suspended to the pubic symphysis and tensioned to allow elevation of the vesicourethral anastomosis. There are four surgeons working at both trial sites who will be involved in performing the radical prostatectomy and sling placement on trial patients. All surgeons have had significant experience in performing radical prostatectomy (> 100 cases each). To ensure sufficient experience in the placement of urethral slings, each surgeon (other than the principle investigator, who has placed over 200 slings) will undergo a training period of 5 patients with sling placement under the proctoring of the principal investigator prior to accrual of the first trial patient from the individual surgeon. All patients will be characterized with respect to age, ethnicity, BMI, prostate size, amount of nerve sparing, preoperative urinary function, surgeon, serum PSA, and tumor characteristics. Prostate size and tumor characteristics will be attained at histological assessment of the prostate specimen by the pathology department. Preoperative urinary function will be assessed by EPIC and IPSS questionnaires at baseline. The amount of nerve sparing will be assessed by the surgeon performing the radical prostatectomy after the prostate dissection is complete. Each side will be assessed separately as complete, partial or no nerve sparing. Stratification will be based upon age at enrollment (<65 years vs. >65 years). For each of the 2 strata patients will be randomized to placement of a sling or not, serving as the control group, on a one to one basis with the assignment determined using a computer software program. Randomization assignment of the planned procedure will be balanced using a fixed block design. Consecutively identified patients undergoing RARP and meeting eligibility criteria for the trial will be approached for involvement in this trial. Patients and study personnel will be blinded as to which patients received slings. Surgeons performing the individual procedures cannot be blinded to the procedure, but will not know the randomization assignment until the prostate dissection is completed and the procedure reaches the stage of sling placement. A sealed envelope containing the randomization assignment of the patient to the sling or non-sling group will be placed at the operating room front desk by the research coordinator prior to the start of surgery. This envelope will not be opened until the prostate is removed. A unique identifying number, that has no association with randomization allocation, will be assigned to each trial patient. These numbers will be placed on envelopes to match them to patients to avoid any confusion on days where multiple trial patients may be undergoing radical prostatectomy. Furthermore, surgeons will not be involved in attaining any outcome data from patients and therefore should not cause any bias to the study outcomes. Investigators expect accrual of 5 patients every week; therefore, investigators estimate that it will take approximately 37 weeks to complete the study accrual of 182 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients undergoing robot assisted radical prostatectomy at UCSF
* Histologically defined adenocarcinoma of the prostate
* English or Spanish speaking patients with the ability to provide informed written consent and willingness to comply with the requirements of the protocol
* Age 40-75 year

Exclusion Criteria:

* · Patients should not have received any radiation or hormonal therapy prior to surgery for any purpose

  * Any prior prostate surgery
  * No current or previous history of urinary incontinence requiring chronic pad use or treatments for urinary incontinence
  * Patients may not be receiving any other investigational agents
  * Any condition that compromises compliance with the objectives and procedures of this protocol, as judged by the principal investigator

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Pad use | 6 months
  The primary objective of this study is to compare the proportion of people requiring 0 pads per day 6 months after RARP in men with and without sling placement. Patients will also be assessed at 1 and 3 months.

SECONDARY OUTCOMES:
Time to zero pads | 6 months
  Determine if there is a difference in median time to continence defined as not requiring any pad post-surgery between those with and without a sling.

OTHER OUTCOMES:
Additional pad use outcomes at one and three months | 3 months
  2.1 Compare the proportion of patients with and without sling placement who use at most 1 pad per day after RARP. Patients will be assessed to determine the frequency at 1, 3 and 6 months.
  2.3 Determine if urinary quality of life as measured by a change from baseline in the Expanded Prostate Cancer Index Composite (EPIC) urinary domain scores differ between sling and non-sling patients at 1, 3 and 6 months 2.4 Determine if urinary obstructive symptoms as measured by a change from baseline in the International Prostate Symptom Score (IPSS) differ between sling and non-sling patients at 1, 3 and 6 months 2.5 Determine if there is a difference in urinary retention at 3 months after surgery between sling and non sling patients.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, San Francisco, California, United States